CLINICAL TRIAL: NCT04974359
Title: Interventional, Randomized, Double-Blind, Crossover, Placebo-Controlled, Multiple-Dose Lu AG06466 Phase IB Study in Patients With Fibromyalgia Using Neuroimaging to Investigate Its Pharmacodynamic Effects on Central Pain Processing and Neuroinflammation
Brief Title: A Study to Evaluate Lu AG06466 in Participants With Fibromyalgia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to enrolment challenges.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19365A
Record Dates: First submitted 2021-06-28; First posted 2021-07-23 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lu AG06466 (Experimental): Participants will receive an oral titrated dose of Lu AG06466 once daily for 22 days in 1 of 2 treatment periods.
  Interventions: Drug: Lu AG06466
- Placebo (Placebo Comparator): Participants will receive an oral dose of placebo matching to Lu AG06466 once daily for 22 days in 1 of 2 treatment periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AG06466 — Lu AG06466 - capsules
  Arms: Lu AG06466
Drug: Placebo — Placebo - capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out the effect of Lu AG06466 on the body in participants with fibromyalgia by assessing pain levels, brain signal changes, and psychiatric (mental) assessments.

DETAILED DESCRIPTION:
This study will include 2 treatment periods and will utilize a crossover study design with a 7- to 14-day washout period between each 22-day treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) of ≥18.5 and ≤38.0 kilograms (kg)/square meter (m^2).
* The participant has a fibromyalgia diagnosis, with self-reported pain visual analogue scale (VAS) score >4, based on a self-reported pain diary assessed for a minimum of 4 out of 7 days prior to the Baseline Visit.
* The participant is, in the opinion of the investigator, eligible based on medical history, a physical examination, a neurological examination, vital signs (including orthostatic vital signs), an electrocardiogram (ECG), and the results of the clinical chemistry, hematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has a disease, including clinically significant liver disease of any origin, or takes medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the study.
* The participant has any other disorder for which the treatment takes priority over the treatment of fibromyalgia in this study or is likely to interfere with the study treatment or impair treatment compliance.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Blood Oxygene Level Dependent (BOLD) Response in the Evoked-Pain Test | Day 22 of each 22-day treatment period
  BOLD response was evaluated using Functional Magnetic Resonance Imaging (fMRI). During the evoked-pain test, each participant will undergo a block design scan, during which 3 cuff pressures ('light touch' = 30 millimeter of mercury [mmHg]; 'equal pressure' = 120 mmHg; 'equal pain' = 40 to 60/100 Numeric Rating Scale [NRS] units) will be applied to the left calf using the pressure cuff device in pseudo random order.
Change in Resting State fMRI (rsfMRI) Functional Connectivity, Assessed by Voxelwise Connectivity Maps Based in Seed Voxels | Day 22 of each 22-day treatment period
  Each participant will undergo a task-free resting state scan, where in they will be instructed to focus on a static fixation cross.
fMRI Data: BOLD Percent Signal Change Under Conditions of Visual Stimulation Versus Fixation | Day 22 of each 22-day treatment period
  Each participant will undergo a block design scan, with alternating blocks of flashing checkerboard and a static fixation cross.

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Collaborative NeuroScience Network LLC, Long Beach, California, United States